CLINICAL TRIAL: NCT03468439
Title: Short Term Effect of Ultrasound and Peripheral Nerve Stimulator Guided Femoral Nerve Block With Phenol on Outcomes in People With Traumatic Spinal Cord Injury
Brief Title: Ultrasound and Peripheral Nerve Stimulator Guided Femoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Principal Investigator, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2018-02-27; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Spinal Cord Injuries
Keywords: nerve block
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Phenol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- femoral nerve block (Other)
  Interventions: Other: Femoral nerve block with phenol

INTERVENTIONS:
Other: Femoral nerve block with phenol

SUMMARY:
A pre-post descriptive study was performed to examine the immediate effects of ultrasound (US) guided femoral nerve block with phenol (UGFNBwP) in managing lower limb spasticity of individuals with traumatic spinal cord injury (SCI).

DETAILED DESCRIPTION:
Study Design: A pre-post descriptive study was performed. Objectives: To examine the immediate effects of ultrasound (US) guided femoral nerve block with phenol (UGFNBwP) in managing lower limb spasticity of individuals with traumatic spinal cord injury (SCI).

Setting: Ankara, Turkey Methods: Nineteen patients with traumatic SCI presenting with lower extremity spasticity were treated with UGFNBwP. Modified Ashworth Scale (MAS) of hip flexion and knee extension, functional independence measure (FIM) motor subscale, difficulty of catheterization (DoC), hygiene score (HS), spasm frequency (SF), sleep quality (SQ) and patient satisfaction (PS) were measured in all patients prior to treatment, at first week and second month.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic etiology
* Duration of spinal cord injury more than twelve months
* Spasticity of hip flexor and/or knee extensor muscle
* Use of any oral medications to reduce spasticity at stable doses for at least one month before first assessment
* The patients have to accept to continue same dose until end of the last assessment
* Medical clearance to participate

Exclusion Criteria:

* Having established contracture of the knee/hip joint
* Aged over 65 years
* History of surgery for knee/hip disorders
* Non-traumatic etiology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | up to 8 weeks
  Scale measures muscle tone (spasticity). (min-max:0-4).Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Functional independence measure | up to 8 weeks
  Scale measures level of independence on activities of daily life (min-max: 0-126) points).Motor subscale of FIM measure is used in this study (min-max:0-91). Higher values represent a better outcome.

IPD SHARING:
Plan to Share IPD: Undecided